CLINICAL TRIAL: NCT00855803
Title: Phase II Study of Stereotactic Body Radiation Therapy and Vertebroplasty for Localized Spinal Metastasis (SBRT Spine)
Brief Title: Stereotactic Body Radiation Therapy and Vertebroplasty in Treating Patients With Localized Spinal Metastasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Robert Timmerman, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 072010-134
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Results first posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-02

CONDITIONS: Metastatic Cancer; Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: spinal cord metastases; unspecified adult solid tumor, protocol specific; pain
MeSH Terms: conditions — Neoplasm Metastasis; Pain | interventions — Radiation; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation followed by Vertebroplasty (Experimental): Intervention:
  This study is one arm. All patients will undergo radiotherapy followed by vertebroplasty. Patients who had prior radiotherapy will undergo 5 fractions of stereotactic body radiotherapy (SBRT) over 30-90 minutes each. Patients has no prior radiotherapy will undergo 1 fraction of SBRT over 30-90 minutes. The full patient population will then undergo vertebroplasty*.
  *Vertebroplasty may not be possible for certain patients due to tumor location or safety. In such cases, patients will omit the vertebroplasty but receive all other protocol care and follow-up.
  Interventions: Radiation: radiation

INTERVENTIONS:
Radiation: radiation — Given in 1 or 5 fractions
  Other Names: stereotactic body radiation therapy

SUMMARY:
RATIONALE: Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Vertebroplasty may help prevent fractures and spinal cord compression caused by spinal metastasis. Giving stereotactic body radiation therapy together with vertebroplasty may help lessen pain and improve quality of life of patients with spinal metastasis.

PURPOSE: This phase II trial is studying how well giving stereotactic body radiation therapy together with vertebroplasty works in treating patients with localized spinal metastasis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy of stereotactic body radiotherapy in reducing pain at 3 months in patients with localized spinal metastasis.

Secondary

* To determine the duration of pain response at the treated site(s) scored as the time of maximal pain relief to an increase of 2 points on the Visual Analogue Scoring System.
* To determine the functional preservation of improvement as measured by the Brief Pain Inventory.
* To prospectively assess quality of life using the FACT-G and EQ-5D questionnaires.
* To determine the long-term stability of the treated vertebral bone (e.g., fracture, sclerotic change, vertebral body height, or malalignment) as measured by MRI, CT scan, and plain radiographs.

OUTLINE: Patients are assigned to 1 of 2 treatment groups according to prior radiotherapy to the planned treatment site(s).

* Group 1 (prior radiotherapy): Patients undergo 5 fractions of stereotactic body radiotherapy (SBRT) over 30-90 minutes each.
* Group 2 (no prior radiotherapy): Patients undergo 1 fraction of SBRT over 30-90 minutes.

Within 1 month after the initiation of SBRT, patients in both groups undergo percutaneous vertebroplasty.

Patients complete pain and quality-of-life questionnaires at baseline and periodically during study. Patients also undergo MRI and CT scan at baseline, at 1, 3, and 6 months, and then every 6 months for 3 years to assess changes in vertebral bone strength and stability.

After completion of study therapy, patients are followed at 2 weeks, at 1, 3, and 6 months, and then every 6 months for 3 years.

ELIGIBILITY:
Eligibility:

Inclusion:

* Patients must have localized spine metastasis (a solitary spine metastasis; two contiguous levels, or up to three separate single vertebral levels are permitted)
* Patients must have a VAS of ≥4 at any of the planned treatment sites
* Patient with epidural, spinal nerve, and/or cord compression on MRI may be included
* Histologic confirmation of cancer is required by biopsy, prior surgery, or re-biopsy
* Narcotic pain prescription and usage information must be available and documented
* Patients must sign study specific consent
* Above the age of 18
* For women of childbearing age a negative pregnancy test is required
* Patients considered for the retreatment arm, must not of had prior radiation to the proposed spinal site within a 3 month interval prior to treatment
* Zubrod score of 0-2

Exclusion:

* Patients who have been non-ambulatory for more than 7 days
* Patients with compression fractures
* Spine instability requiring fixation
* Patients with paraspinal extension
* Patients with bony fragments
* Planned systemic treatment within one week after treatment.
* Absence of pathological diagnosis of cancer
* Chemotherapy within one week of treatment
* Patients with Multiple Myeloma, Lymphoma, or Plasmacytoma
* Patient suffered from unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
* Patient had a transmural myocardial infarction within the last 6 months
* Patient has an acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
* Patient has hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
* PT is not within normal limits or planned and feasible to be corrected to normal limits prior to vertebroplasy
* PTT is not within normal limits or planned and feasible to be corrected to normal limits prior to vertebroplasy
* Platelet count is < 50,000
* History of significant psychiatric illness

Note: Vertebroplasty may not be possible for certain patients due to tumor location or safety. In such cases, patients will omit the vertebroplasty but receive all other protocol care and follow-up Visual Analog Scoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-02; Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Timmerman, MD, Principal Investigator — Simmons Cancer Center
Locations (1):
- University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 withdrew before starting treatment, 1 had clinical decline prior to treatment and was removed, 1 was removed prior to treatment for local progression, and 1 was removed due to a pre-existing compression fracture prior to treatment, These 6 patients did start the study but were assessed for other outcomes.
Groups:
- Total Population: All patients enrolled to the study
Period: Overall Study
Arm/Group | Total Population
Started | 35
Completed | 21
Not Completed | 14
Not completed — Death | 2
Not completed — Lost to Follow-up | 2
Not completed — Technical inability to undergo procedure | 2
Not completed — Not evaluable at 3 month timepoint | 2
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: 35 patients enrolled to the study, 29 patients started protocol treatment and had study specific measures completed.
Arm/Group | Total Population
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 60 [40 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Primary Site [Number; unit: participants] — Population: 35 patients enrolled to the study, 29 patients started protocol treatment and had study specific measures completed.
  participants
    Lung: number analyzed (Participants) | 29
    Lung | 10
    Breast: number analyzed (Participants) | 29
    Breast | 4
    Prostate: number analyzed (Participants) | 29
    Prostate | 4
    Kidney: number analyzed (Participants) | 29
    Kidney | 4
    Melanoma: number analyzed (Participants) | 29
    Melanoma | 3
    Colorectal: number analyzed (Participants) | 29
    Colorectal | 2
    Oropharyngeal: number analyzed (Participants) | 29
    Oropharyngeal | 1
    Thyroid: number analyzed (Participants) | 29
    Thyroid | 1
Spine Location [Number; unit: participants] — Population: 35 patients enrolled to the study, 29 patients started protocol treatment and had study specific measures completed.
  participants
    Cervical: number analyzed (Participants) | 29
    Cervical | 4
    Thoracic: number analyzed (Participants) | 29
    Thoracic | 12
    Lumbar: number analyzed (Participants) | 29
    Lumbar | 13
Number of vertebrae treated [Number; unit: participants] — Population: 35 patients enrolled to the study, 29 patients started protocol treatment and had study specific measures completed.
  participants
    1: number analyzed (Participants) | 29
    1 | 23
    2: number analyzed (Participants) | 29
    2 | 6
Preexisting endplate fracture [Number; unit: participants] — Population: 35 patients enrolled to the study, 29 patients started protocol treatment and had study specific measures completed.
  participants
    Yes: number analyzed (Participants) | 29
    Yes | 5
    No: number analyzed (Participants) | 29
    No | 24

OUTCOME MEASURES:

1. Primary Outcome: Pain Response as Measured by VAS at 3 Months
Description: Pain reduction as measured by Visual Analogue Scoring System (VAS) at 3 months
  Patient pain was recorded on a 10-point scale (0: no pain, 10: most severe pain). At baseline patients were required to have a pain score of 4 or higher associated with spine metastases. Pain response was recorded again during follow-up visits to determine the pain response:
  A pain score of 0 represents a complete response A decrease in the pain score by at least 2 points represents a partial response VAS scores were used to determine the number of patients with a partial pain response, with a complete pain response, and without a pain response
Time Frame: 3 month
Population: Patients who were evaluable at the 3-month timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Total Population
Number analyzed (Participants) | 21
Participants
  Patients with a partial pain response at 3 months | 8
  Patients with a complete pain response at 3 months | 12
  Patients without a pain response | 1

2. Secondary Outcome: Pain Response
Description: Duration of pain response as measured by VAS at 1 month
  Patient pain was recorded on a 10-point scale (0: no pain, 10: most severe pain). At baseline patients were required to have a pain score of 4 or higher associated with spine metastases. Pain response was recorded again during follow-up visits to determine the pain response:
  A pain score of 0 represents a complete response A decrease in the pain score by at least 2 points represents a partial response VAS scores were used to determine the number of patients with a partial pain response, with a complete pain response, and without a pain response
Time Frame: 1 month
Population: Patients who were evaluable at the 1 month timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Total Population
Number analyzed (Participants) | 25
Participants
  Patients with a complete pain response | 10
  Patients with a partial pain response | 10
  Patients with no pain response | 5

3. Secondary Outcome: Overall Survival
Description: Overall survival measured from the date of accession to the date of death. Median times will be reported.
Time Frame: 5 year
Population: Patients who received spine SABR
Measure: Median (Full Range); unit: months
Arm/Group | Total Population
Number analyzed (Participants) | 29
months | 9 [0 to 63.4]

4. Secondary Outcome: Daily Function
Description: Time to functional decline as measure by the Brief Pain Inventory (BPI) at baseline. BPI has two sections that are scored- pain severity and pain interference. For each of these a numeric scale from 0-10 is used, with 0 being the worst pain and 10 being the worst pain.
Time Frame: Baseline
Population: Patients enrolled to the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Population
Number analyzed (Participants) | 35
score on a scale
  Pain Severity | 5.8 (1.8)
  Pain Interference | 6.0 (2.2)

5. Secondary Outcome: Quality of Life Questionnaire Responses
Description: Number of participants who filled out the Functional Assessment of Cancer Therapy- General (FACT-G) and the European Quality of Life Five Dimension (EQ-5D) questionnaires at baseline, 1, 3, 6, and 12 months
Time Frame: 12 months
Population: Enrolled participants
Measure: Number; unit: participant responses
Arm/Group | Total Population
Number analyzed (Participants) | 35
participant responses
  Number of responses at baseline | 35
  Number of responses at 1 month | 29
  Number of responses at 3 months | 21
  Number of responses at 6 months | 16
  Number of responses at 12 months | 7

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Total Population
All-Cause Mortality (participants affected / at risk) | 2/29
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 3/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Population (N=29)
Acute myelopathy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Population (N=29)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Acute hematoma (Injury, poisoning and procedural complications) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Metastatic renal cell carcinoma (Renal and urinary disorders) | 1 (1)
Spinal canal stenosis (Nervous system disorders) | 1 (1)
Laminectomy (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT00855803/Prot_SAP_000.pdf